CLINICAL TRIAL: NCT02962154
Title: Neurocardiac Interactions Evaluated by Anatomic and Physiologic MRI Assessment
Acronym: NIRVANA
Status: Withdrawn | Type: Observational
Why Stopped: Our physician researcher left WCM after the trial was approved.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1405015093
Record Dates: First submitted 2015-04-20; First posted 2016-11-11 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Ischemia; Stress, Mental
Keywords: Invasive Coronary Angiography; Myocardial Infarction; Major Depressive Disorder; Bipolar I Disorder; Bipolar II Disorder; Mental Stress
MeSH Terms: conditions — Ischemia; Stress, Psychological; Myocardial Infarction; Depressive Disorder, Major; Bipolar Disorder | interventions — Health Status; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2mL of blood will be drawn for sample banking for future research studies ONLY from subjects who provide permission for storing their sample for use in future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Coronary Artery Disease (CAD): Patients with known coronary artery disease (CAD) as defined by prior PCI, CABG, prior MI, prior abnormal stress test, or invasive coronary angiography (ICA) and who are hemodynamically stable
  They will undergo the following:
  Radiation: Coronary CT Angiography Other: Mood Symptom Scale Other: Anxiety Symptom Scale Other: Chronic Stress Inventories Other: Psychosocial Function Questionnaires Other: General Health and quality of life questionnaires Other: Magnetic Resonance Imaging
  Interventions: Radiation: Coronary CT Angiography; Other: Mood Symptom Scale; Other: Anxiety Symptom Scale; Other: Chronic Stress Inventories; Other: Psychosocial Function Questionnaires; Other: General Health and quality of life questionnaires; Other: Magnetic Resonance Imaging
- Major Depressive Disorder: Patients with a diagnosis of major depressive disorder and/or a diagnosis of bipolar 1 or bipolar 2 disorder
  They will undergo the following:
  Radiation: Coronary CT Angiography Other: Mood Symptom Scale Other: Anxiety Symptom Scale Other: Chronic Stress Inventories Other: Psychosocial Function Questionnaires Other: General Health and quality of life questionnaires Other: Magnetic Resonance Imaging
  Interventions: Radiation: Coronary CT Angiography; Other: Mood Symptom Scale; Other: Anxiety Symptom Scale; Other: Chronic Stress Inventories; Other: Psychosocial Function Questionnaires; Other: General Health and quality of life questionnaires; Other: Magnetic Resonance Imaging

INTERVENTIONS:
Radiation: Coronary CT Angiography — The coronary CT angiography will assess for coronary artery stenosis, plaque characteristics, calcifications, and other factors.
Other: Mood Symptom Scale — Some or all of the following questionnaires will be conducted to assess mood symptoms:
  Beck Depression Inventory, Hamilton Depression Rating Scale (24-item), Montgomery Asberg Depression Rating Scale (MADRS), Mood and Anxiety Symptom Questionnaire (MASQ), QIDS, Young Mania Rating Scale
Other: Anxiety Symptom Scale — Some or all of the following questionnaires will be conducted to assess anxiety symptoms:
  Beck Anxiety Inventory, Spielberger State/Trait Anxiety Inventory (STAI), GAD-7 Anxiety Questionnaire, Penn State Worry Questionnaire (PSWQ)
Other: Chronic Stress Inventories — Some of all of the following questionnaires will be conducted to assess chronic stress:
  Chronic stress inventories: Cohen Perceived Stress Scale, Holmes and Rahe Stressful Life Events Scale, Karasek Job Strain Questionnaire, Conner-Davidson Resilience Scale, PTSD Checklist
Other: Psychosocial Function Questionnaires — Some of all of the following questionnaires will be conducted to assess psychosocial function:
  Type A Personality Scale, NEO Personality Inventory, Positive and Negative Affect Schedule (PANAS), Behavioral Inhibition/Behavioral Approach Scale (BIS/BAS)
Other: General Health and quality of life questionnaires — Some of all of the following questionnaires will be conducted to assess quality of life:
  EQ-5D Health Questionnaire, Seattle Angina Questionnaire, International Index of Erectile Function (ILEF-5), Pittsburgh Sleep Quality Scale, Morningness Eveningness Questionnaire
Other: Magnetic Resonance Imaging — First, subjects will undergo a resting cardiac MR perfusion study to establish baseline (pre-stress) measures of cardiovascular function. Second, subjects will undergo a series of brain magnetic resonance imaging studies (T1-weighted anatomical MRI, diffusion tensor imaging, resting state functional MRI) to establish baseline (pre-stress) measures of brain function and structural correlates. Third, investigators will use a well-validated cognitive task to induce mental stress by testing subjects' working memory for a series of emotionally arousing or neutral images, while repeating the functional MRI scan. Finally, subjects will undergo a repeat cardiac MR perfusion study while being tested on the same mental stress task.

SUMMARY:
The purpose of project is to answer fundamental questions about the mechanisms underlying mental stress ischemia in patients with coronary artery disease, mood disorders, or both, and to identify potential biomarkers and psychosocial risk factors associated with this condition.

To achieve this goal, investigators will use cutting-edge cardiovascular and functional neuroimaging tools to study mental stress ischemia in a carefully controlled laboratory setting in subjects recruited from four patient populations: 1) patients who recently sustained a myocardial infarction; 2) patients undergoing non-emergent invasive coronary angiography (with and without known coronary artery disease); 3) patients with a diagnosis of major depressive disorder; and 4) patients with a diagnosis of bipolar 1 or bipolar 2 disorder.

DETAILED DESCRIPTION:
Mental stress ischemia occurs when a psychosocial or mental stressor triggers an imbalance between the supply and demand for oxygen by cardiac myocytes. Epidemiological studies indicate that mental stress ischemia is common, occurring in 20-25% of patients with coronary artery disease (CAD) and portends a poor prognosis. The underlying mechanisms are thought to involve stress-induced activation of the sympathetic nervous system and associated effects on cardiovascular function. But how neurobiological and cardiovascular factors interact to generate mental stress ischemia is unknown. Furthermore, patients with major depressive disorder, bipolar disorder, and other stress-related psychiatric conditions have elevated rates of cardiovascular co-morbidities, including sudden cardiac death, yet mental stress ischemia has not been studied extensively in these psychiatric populations. The purpose of project is to answer fundamental questions about the mechanisms underlying mental stress ischemia in patients with coronary artery disease, mood disorders, or both, and to identify potential biomarkers and psychosocial risk factors associated with this condition.

To achieve this goal, investigators will use cutting-edge cardiovascular and functional neuroimaging tools to study mental stress ischemia in a carefully controlled laboratory setting in subjects recruited from four patient populations: 1) patients who recently sustained a myocardial infarction; 2) patients undergoing non-emergent invasive coronary angiography (with and without known coronary artery disease); 3) patients with a diagnosis of major depressive disorder; and 4) patients with a diagnosis of bipolar 1 or bipolar 2 disorder.

ELIGIBILITY:
Inclusion Criteria for Cardiac Subjects:

1. Male and female subjects, ages 50 years or more
2. Able to provide informed consent. Must be fluent english speakers.
3. Known coronary artery disease (CAD) as defined by prior PCI, CABG, prior MI, prior abnormal stress test or invasive coronary angiography (ICA)
4. Patients that are hemodynamically stable

Exclusion Criteria for Cardiac subjects:

1. Evidence of ongoing myocardial infarction or homonymic instability
2. Positive pregnancy test or unknown pregnant state at the time of enrollment for all women of child-bearing potential
3. Known contraindications to cardiovascular CT angiography with intravenous contrast (A) Known allergies (B) Renal dysfunction (GFR < 30ml/min) (C) Contraindications to beta-blockers or nitroglycerin or adenosine (D) Irregular heart rate not controlled by administration of beta-blockers
4. Patients with contraindications to MRI scans (A) Non-MR compatible device or material implant (B) Known allergies to gadolinium containing contrast agent (C) Renal dysfunction (GFR < 30 ml/min)

Inclusion Criteria for Psychiatric Subjects

1. Male and female subjects, ages 50 years or more
2. Must be fluent English-speakers due to the design of the mental stress tasks. Able to provide informed consent.
3. Subjects who are stable and meet DSM-V criteria for a diagnosis of major depressive disorder, bipolar 1 disorder, or bipolar 2 disorder, as assessed in an initial screening interview by phone and confirmed by a structured clinical interview on the first day of the study.

Exclusion Criteria for Psychiatric Subjects:

1. Subjects with a history of seizure disorder, stroke, Parkinson's disease, any form of dementia, or head injury resulting in loss of consciousness will be excluded from this study.
2. Contraindications to MRI be assessed during the screening interview and again using the NY-Presbyterian Hospital MRI Checklist prior to scanning and will also serve as exclusion criteria. They include claustrophobia; a history of metal implants (including braces, orthopedic implant, cochlear implant, implanted cardiac pacemaker, implanted cardioverter defibrillator, and ocular implant); weight over 250 pounds (owing to the size of the MR scanner bore); and women who are currently pregnant or breastfeeding.
3. Subjects who indicate that there is a chance that they may be pregnant will be asked to take a pregnancy test. They will be informed of the potential for false positive results due to diet, vitamins, and supplements, or over-the-counter medications. A positive pregnancy test will necessitate exclusion from the study, and the results will be disclosed to the participant.
4. Patients who are currently being treated with a beta blocker or daily (standing) benzodiazepines will be excluded, unless, in the judgment of the prescribing physician, the dose can be withheld on the morning of the each study session, due to the potential for these medications to mask neurobiological and cardiovascular responses to mental stress.
5. Investigators will also assess for additional psychiatric exclusion criteria during the screening interview and structured clinical interview: patients with bipolar 1 disorder who are currently manic; patients with any mood disorder currently complicated by hallucinations, delusions, or other psychotic features; patients with active suicidal ideation; and patients meeting DSM-V criteria for a co-morbid substance abuse disorder within the last 12 months will all be excluded. Other psychiatric co-morbidities will be permitted.

Subjects who meet both the psychiatric and cardiac inclusion criteria will also be enrolled in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll male and female subjects 50 years of age or older who have:
  1. recently sustained a myocardial infarction
  2. undergone or are undergoing non-emergent invasive coronary angiography (with and without known coronary artery disease)
  3. a diagnosis of major depressive disorder; and a diagnosis of bipolar 1 or bipolar 2 disorder
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mental stress induced ischemia as measured by cardiac MRI | 2 weeks
  Subjects will undergo a brief training program for low-stress version of emotion regulation task and working memory task on a laptop. Baseline (non-stress) resting cardiac MR perfusion and baseline (non-stress) brain MRI studies. In addition to a mental stress task brain fMRI and mental stress cardiac MR perfusion. We can analyze the prevalence of mental stress induced ischemia.

SECONDARY OUTCOMES:
Change in cardiac stress perfusion as measured by cardiac MRI (pre and post mental stress) | 2 weeks
  We will test for within-subject changes in cardiovascular function and neural activity in stress-sensitive brain circuits, comparing pre and post-stress cardiac mRI and brain MRI studies.

CONTACTS AND LOCATIONS:
Overall Officials: James K Min, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided